CLINICAL TRIAL: NCT00129389
Title: Multicenter Randomized Phase III Trial to Compare 6 FAC Cycles vs 4 FAC Cycles Followed by 8 Weekly Paclitaxel Administrations, as Adjuvant Treatment for Node Negative Operable Breast Cancer Patients
Brief Title: FAC Versus FAC Plus Weekly Paclitaxel as Adjuvant Treatment of Node Negative High Risk Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM 2003-02; 2005-003109-10 (EudraCT Number)
Record Dates: First submitted 2005-08-10; First posted 2005-08-11 (Estimated); Results first posted 2019-07-12 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: Node negative, high risk breast cancer.; Prognostic gene profile.; Saint Gallen high risk criteria.; Weekly paclitaxel.
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Doxorubicin; liposomal doxorubicin; Cyclophosphamide; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: FAC (Active Comparator): FAC X 6 The standard arm consisted of six cycles of FAC (fluorouracil 500 mg/m2, doxorubicin 50mg/m2, and cyclophosphamide 500mg/m2) administered once every 3 weeks.
  Interventions: Drug: Fluorouracil; Drug: Doxorubicin; Drug: Cyclophosphamide
- Arm B: FAC-wP (Experimental): FAC X 4 + 8 weekly Paclitaxel (wP) Patients in the experimental arm received four cycles of the FAC regimen followed by eight weekly administrations of paclitaxel (100mg/m2 per dose)
  Interventions: Drug: Fluorouracil; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Paclitaxel

INTERVENTIONS:
Drug: Fluorouracil — Arm A: FAC Arm B: FAC-wP
  Other Names: Adrucil
Drug: Doxorubicin — Arm A: FAC Arm B: FAC-wP
  Other Names: Caelyx
Drug: Cyclophosphamide — Arm A: FAC Arm B: FAC-wP
  Other Names: Cytoxan
Drug: Paclitaxel — Arm B: FAC-wP
  Other Names: taxol
  Arms: Arm B: FAC-wP

SUMMARY:
This is a prospective, open-label, randomized, phase III trial. Patients will be stratified after breast surgery, as per investigational site; menopausal status; node negative diagnosis, as per sentinel-node technique versus lymphadenectomy; hormone receptor status (positive versus negative).

DETAILED DESCRIPTION:
Patients will be randomized to:

* Fluorouracil, doxorubicin, and cyclophosphamide (FAC) x 6 (cycles): 5-fluorouracil 500 mg/m2 + doxorubicin 50 mg/m2 + cyclophosphamide 500 mg/m2 day 1, every 3 weeks, for 6 cycles.
* FAC x 4 (cycles) → Paclitaxel x 8 (cycles): 5-fluorouracil 500 mg/m2 + doxorubicin 50 mg/m2 + cyclophosphamide 500 mg/m2 day 1, every 3 weeks, for 4 cycles, followed by 8 administrations of weekly paclitaxel 100 mg/m2

Premenopausal women with hormone receptor positive tumors must receive tamoxifen 20 mg daily for 5 years, after the end of chemotherapy.

Postmenopausal women with hormone receptor positive tumors are allowed to receive aromatase inhibitors as initial adjuvant hormone therapy or after tamoxifen.

All patients with breast conservative surgery must receive radiotherapy.

Estimated 5-year disease-free survival in the control arm (FAC x 6) is expected to be 80%. It is expected that disease-free survival will increase by 5% in the experimental arm (FAC-paclitaxel). 906 patients per arm must be recruited, to detect this difference with an alpha error of 0.05 and 80% power. Assuming a 6% post-randomization drop-out rate, 960 patients per arm are needed, 1920 in total.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Histological diagnoses of operable invasive adenocarcinoma of the breast (T1-T3). Tumors must be Human Epidermal Growth Factor Receptor 2 (HER2) negative. Patients must be free of disease in the axilla (node negative). If lymphadenectomy is done, at least 10 nodes must be examined. If sentinel node technique is used, sentinel node must be free of disease. Patients must present at least one high risk criterion (St. Gallen, 1998) as follows:

  * Tumor size > 2 cm; and/or
  * ER and Progesterone Receptor (PgR) negative; and/or
  * Histological grade 2-3; and/or
  * Age < 35 years old.
* Time window between surgery and study randomization must be less than 60 days.
* Surgery must consist of mastectomy or conservative surgery. Margins free of disease and ductal carcinoma in situ (DCIS) are required. Lobular carcinoma is not considered a positive margin.
* Patients must not present evidence of metastatic disease.
* Status of hormone receptors in primary tumor. Results must be available before the end of adjuvant chemotherapy.
* Status of HER2 in primary tumor, known before randomization. Patients with Immunohistochemistry (IHC) 0 or +1 are eligible. For patients with IHC 2+, fluorescent in situ hybridization (FISH) is mandatory and result must be negative.
* Age >= 18 and <= 70 years old.
* Performance status (Karnofsky index) >= 80.
* Normal electrocardiogram (EKG) in the 12 weeks prior to randomization. If needed, normal cardiac function must be confirmed by left ventricular ejection fraction (LVEF).
* Laboratory results (within 14 days prior to randomization):

  * Hematology: neutrophils >= 1.5 x 10^9/l; platelets >= 100x 10^9/l; hemoglobin >= 10 mg/dl;
  * Hepatic function: total bilirubin <= 1 upper normal limit (UNL); Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) <= 2.5 UNL; alkaline phosphatase <= 2.5 UNL. If values of AST and ALT > 1.5 UNL are associated with alkaline phosphatase > 2.5 UNL, patient is not eligible.
  * Renal function: creatinine <= 175 mmol/l (2 mg/dl); creatinine clearance >= 60 ml/min.
* Complete stage workup during the 12 weeks prior to randomization (mammograms are allowed within a 20 week time window). All patients must have a bilateral mammogram, thorax x-ray, abdominal echography and/or computed tomography (CT)-scan. If bone pain, and/or alkaline phosphatase elevation, a bone scintigraphy is mandatory. This test is recommended for all patients. Other tests, as clinically indicated.
* Patients able to comply with treatment and study follow-up.
* Negative pregnancy test done in the 14 previous days to randomization.

Exclusion Criteria:

* Prior systemic therapy for breast cancer.
* Prior therapy with anthracyclines or taxanes (paclitaxel or docetaxel) for any malignancy.
* Prior radiotherapy for breast cancer.
* Bilateral invasive breast cancer.
* Pregnant or lactating women. Adequate contraceptive methods must be used during chemotherapy and hormone therapy treatments. Negative pregnancy test in the 14 previous days to randomization.
* Any T4 or N1-3 or M1 tumor.
* HER2 positive breast cancer (IHC 3+ or positive FISH result).
* Pre-existing grade >=2 motor or sensorial neurotoxicity by the National Cancer Institute Common Toxicity Criteria (NCICTC) v-2.0.
* Any other serious medical pathology, such as congestive heart failure, unstable angina, history of myocardial infarction during the previous year, uncontrolled hypertension or high risk arrhythmias.
* History of neurological or psychiatric disorders, which could preclude the patients to free informed consent.
* Active uncontrolled infection.
* Active peptic ulcer; unstable diabetes mellitus.
* Previous or current history of neoplasms different from breast cancer, except for skin carcinoma, cervical in situ carcinoma, or any other tumor curatively treated and without recurrence in the last 10 years; ductal in situ carcinoma in the same breast; lobular in situ carcinoma.
* Concomitant treatment with other investigational products. Participation in other clinical trials with a non-marketed drug in the 20 previous days before randomization.
* Concomitant treatment with other therapy for cancer.
* Males.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1925 (Actual)
Dates: Start 2003-09-19 (Actual); Primary Completion 2013-10-01 (Actual); Study Completion 2013-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Universitario San Carlos
Locations (68):
- Spain (68):
  - Hospital General Univ. De Elche, Elche, Alicante
  - Hospital General de Elda, Elda, Alicante
  - Complejo Hospitalario de Manresa, Manresa, Barcelona
  - Consorci Sanitari Parc Tauli, Sabadell, Barcelona
  - Hospital del Espíritu Santo, Santa Coloma de Gramenet, Barcelona
  - Consorci Sanitari Terrassa, Terrassa, Barcelona
  - Hospital Mutua Terrassa, Terrassa, Barcelona
  - Hospital General Jerez de la Frontera, Jerez de la Frontera, Cadiz
  - Hospital Provincial de Castellón, Castellon, Castellón
  - Hospital Comarcal de Barbastro, Barbastro, Huesca
  - Hospital Insular de Gran Canaria, Las Palmas de Gran Canaria, Las Palmas
  - Fundación Hospital de Alcorcón, Alcorcón, Madrid
  - Hospital Madrid- Montepríncipe, Boadilla del Monte, Madrid
  - Hospital de Móstoles, Móstoles, Madrid
  - Hospital Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Policlínico Vigo POVISA, Vigo, Pontevedra
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Sant Joan de Reus, Reus, Tarragona
  - Hospital de la Ribera, Alzira, Valencia
  - Complejo Hospitalario Juan Canalejo, A Coruña
  - Centro Oncológico de Galicia, A Coruña
  - Complejo Hospitalario de Albacete, Albacete
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Virgen de los Lirios, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Clínica Corochan S.A., Barcelona
  - Hospital Clinic i Provincial, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital General de Vic, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital General Yagüe, Burgos
  - Hospital Puerta del Mar, Cadiz
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital Reina Sofía, Córdoba
  - Hospital Virgen de la Luz, Cuenca
  - ICO Hospital Universitari Josep Trueta, Girona
  - Hospital General de Guadalajara, Guadalajara
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Xeral Calde, Lugo
  - Hospital Universitario La Princesa, Madrid
  - Hospital Doce de Octubre, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Ruber Internacional, Madrid
  - Hospital Puerta de Hierro, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital La Paz, Madrid
  - CIOCC Hospital Norte-Sanchinarro, Madrid
  - Complejo Hospitalario Virgen de la Victoria, Málaga
  - Hospital Carlos Haya, Málaga
  - Hospital Morales Messeguer, Murcia
  - Hospital Sta María Nai, Ourense
  - Hospital General Río Carrión, Palencia
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Instituto Oncológico de Guipuzcoa, San Sebastián
  - Hospital de Donostia, San Sebastián
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Univ. Virgen del Rocío, Seville
  - Hospital Universitario de Valme, Seville
  - Hospital Virgen de la Salud, Toledo
  - Hospital Universitario La Fe, Valencia
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital Provincial de Zamora, Zamora
  - Hospital Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Result] Martin M, Ruiz A, Ruiz Borrego M, Barnadas A, Gonzalez S, Calvo L, Margeli Vila M, Anton A, Rodriguez-Lescure A, Segui-Palmer MA, Munoz-Mateu M, Dorca Ribugent J, Lopez-Vega JM, Jara C, Espinosa E, Mendiola Fernandez C, Andres R, Ribelles N, Plazaola A, Sanchez-Rovira P, Salvador Bofill J, Crespo C, Carabantes FJ, Servitja S, Chacon JI, Rodriguez CA, Hernando B, Alvarez I, Carrasco E, Lluch A. Fluorouracil, doxorubicin, and cyclophosphamide (FAC) versus FAC followed by weekly paclitaxel as adjuvant therapy for high-risk, node-negative breast cancer: results from the GEICAM/2003-02 study. J Clin Oncol. 2013 Jul 10;31(20):2593-9. doi: 10.1200/JCO.2012.46.9841. Epub 2013 Jun 3. PMID 23733779
- See also: Spanish Breast Cancer Research Group (GEICAM) is a Spanish Breast Cancer Research Group — http://www.geicam.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1925 patients from 67 Spanish sites were assigned to receive FAC-wP (n=951) or FAC (n=974). 8 patients received no treatment (5 FAC-wP, 3 FAC), and 17 were not treated with the study medication to which they were randomly assigned (1 FAC, 16 FAC-wP). A total of 1,917 patients were evaluable for safety (931 FAC-wP, 986 FAC).
Period: Overall Study
Arm/Group | Arm A: FAC | Arm B: FAC-wP
Started | 974 | 951
Completed | 941 (1 patient was crossed from arm A to B by error. 16 patients were crossed from arm B, to A by error.) | 811 (16 patients were crossed from arm B to A by error. 1 patient was crossed from arm A to B by error.)
Not Completed | 33 | 140
Not completed — Adverse Event | 19 | 87
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 0 | 4
Not completed — Protocol Violation | 0 | 6
Not completed — Withdrawal by Subject | 9 | 23
Not completed — Relapse | 1 | 0
Not completed — Not eligible | 1 | 2
Not completed — Crossed to the other arm | 1 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: FAC | Arm B: FAC-wP | Total
Number analyzed (Participants) | 974 | 951 | 1925
Age, Continuous [Median (Full Range); unit: years] | 50.95 [24 to 75] | 50.89 [24 to 72] | 50.92 [24 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 974 | 951 | 1925
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 960 | 935 | 1895
  Oriental | 3 | 0 | 3
  Hispanic | 10 | 12 | 22
  Other | 1 | 4 | 5
Karnofsky Performance Status (PS) [Count of Participants; unit: Participants] — The Karnofsky PS Index classify patients as to their functional impairment. The lower the Karnofsky score, the worse the survival.
  100 to 80: Able to carry on normal activity and to work; no special care needed.
  70 to 50: Unable to work; able to live at home and care for most personal needs; varying amount of assistance needed.
  40 to 0: Unable to care for self; requires equivalent of institutional or hospital care; disease may be progressing rapidly.
  Participants
    PS 80 | 8 | 7 | 15
    PS 90 | 91 | 81 | 172
    PS 100 | 873 | 863 | 1736
    Not done | 2 | 0 | 2
Menopausal status [Count of Participants; unit: Participants]
  Premenopausal | 472 | 482 | 954
  Peri/postmenopausal | 502 | 469 | 971
Tumor size [Count of Participants; unit: Participants] — Tumor (T) size describes the size of the tumour. Larger T is associated with inferior survival.
  TX: can't be assessed. Tis: ductal carcinoma in situ. T1: tumour is 2 centimetres (cm) across or less. T1mi: tumour is 0.1cm across or less T1a: tumour >0.1 cm but <0.5 cm T1b: tumour >0.5 cm but <1 cm T1c: tumour >1 cm but <2 cm T2: tumour >2 cm but <5 cm across. T3: tumour >5 cm across. T4a: tumour has spread into the chest wall T4b: tumour has spread into the skin and the breast might be swollen T4c: tumour has spread to both the skin and the chest wall T4d: inflammatory carcinoma
  Participants
    T1 | 557 | 569 | 1126
    T2 | 403 | 369 | 772
    T3 | 14 | 13 | 27
Histologic type [Count of Participants; unit: Participants]
  Invasive Ductal Carcinoma | 832 | 813 | 1645
  Invasive Lobular Carcinoma | 71 | 89 | 160
  Other | 71 | 49 | 120
Histologic grade [Count of Participants; unit: Participants] — Cancer cells are given a Grade (G) when they are removed from the breast and checked under a microscope. The G is based on how much the cancer cells look like normal cells.
  G1 or well differentiated (score 3, 4, or 5): cells are slower-growing, and look more like normal breast tissue.
  G2 or moderately differentiated (score 6, 7): cells are growing at a speed of and look like cells somewhere between G1 and 3.
  G3 or poorly differentiated (score 8, 9): cells look very different from normal and will probably grow and spread faster.
  Participants
    GX: Differenciation cannot be assessed | 35 | 36 | 71
    G1: Well differenciated | 64 | 61 | 125
    G2: Moderately differenciated | 446 | 434 | 880
    G3: Poorly differenciated | 429 | 420 | 849
Hormonal receptors [Count of Participants; unit: Participants]
  ER positive and/or PR positive | 713 | 693 | 1406
  ER negative and/or PR negative | 261 | 258 | 519
Human Epidermal growth factor Receptor 2 (HER2) status [Count of Participants; unit: Participants]
  HER2 positive | 95 | 86 | 181
  HER2 negative | 858 | 846 | 1704
  Unknown | 21 | 19 | 40
Triple-negative disease [Count of Participants; unit: Participants]
  Triple-negative disease | 218 | 224 | 442
  Non triple-negative disease | 735 | 708 | 1443
  Unknown | 21 | 19 | 40
Type of surgery [Count of Participants; unit: Participants]
  Mastectomy | 261 | 265 | 526
  Conservative | 713 | 686 | 1399
Axillary surgery [Count of Participants; unit: Participants]
  Lymphadenectomy | 559 | 551 | 1110
  Sentinel node biopsy | 402 | 384 | 786
  Lymphadenectomy + Sentinel node biopsy | 13 | 16 | 29

OUTCOME MEASURES:

1. Primary Outcome: Disease-free Survival (DFS) Event
Description: DFS is defined as the evidence of local, regional or metastatic recurrence, second primary cancer (with the exception of carcinoma of squamous cells or basal cells of the skin, cervical carcinoma in situ or lobular or ductal carcinoma in situ of the breast) or death for any reason.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: FAC | Arm B: FAC-wP
Number analyzed (Participants) | 974 | 951
Participants | 98 | 71

2. Secondary Outcome: Overall Survival (OS) Event
Description: OS event is defined as the death from any cause.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: FAC | Arm B: FAC-wP
Number analyzed (Participants) | 974 | 951
Participants | 40 | 31

ADVERSE EVENTS:
Time Frame: Through study treatment up to 30 days after last study dose; All-Cause Mortality was assessed up to 5 years.
Description: Only Adverse Events grade 3 and 4 were collected. All Serious Adverse Events (SAEs) grade 1, 2, 3, 4 and 5 were collected.
Arm/Group | Arm A: FAC | Arm B: FAC-wP
All-Cause Mortality (participants affected / at risk) | 40/974 | 31/951
Serious Adverse Events (participants affected / at risk) | 60/974 | 61/951
Other Adverse Events (participants affected / at risk) | 442/974 | 523/951
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: FAC (N=974) | Arm B: FAC-wP (N=951)
Febrile neutropenia (Blood and lymphatic system disorders) | 31 | 18 — Grade 3
Neutropenia (Blood and lymphatic system disorders) | 6 | 1 — Grade 4
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 5 | 3 — Grade 3 or 4
Infection without neutropenia (Infections and infestations) | 2 | 6 — Grade 3
Neutropenia (Blood and lymphatic system disorders) | 3 | 1 — Grade 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 — Grade 2
Vomiting (Gastrointestinal disorders) | 1 | 2 — Grade 3
Catheter-related infection (Skin and subcutaneous tissue disorders) | 1 | 1 — Grade 3
Wound-infectious (Infections and infestations) | 1 | 0 — Grade 3
Thrombosis/embolism (Cardiac disorders) | 1 | 3 — Grade 3
CNS cerebrovascular ischemia (Nervous system disorders) | 1 | 0 — Grade 4
Fistula-rectal/anal (Gastrointestinal disorders) | 1 | 0 — Grade 4
Hepatic - Hepatitis (Hepatobiliary disorders) | 1 | 0 — Grade 3
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 | 0 — Grade 2
Diarrhea (Gastrointestinal disorders) | 0 | 2 — Grade 2
Constipation (Gastrointestinal disorders) | 0 | 1 — Grade 3
Gastroenteritis (Gastrointestinal disorders) | 0 | 1 — Grade 2
Vomiting (Gastrointestinal disorders) | 0 | 1 — Grade 2
Gastrointestinal - appendicitis surgery (Gastrointestinal disorders) | 0 | 1
Bone Fracture (General disorders) | 0 | 1 — Grade 3
Pneumonitis, refractory septic shock (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Grade 4
Dizziness (Nervous system disorders) | 0 | 1 — Grade 2
Neurotoxicity (Nervous system disorders) | 0 | 1 — Grade 3
Thrombosis/embolism (Cardiac disorders) | 0 | 3 — Grade 4
Musculoskeletal - Right Essential Coxoartrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Grade 3
Hyperglycemia (Investigations) | 0 | 1 — Grade 3
Fever (General disorders) | 2 | 2 — Grade 1
Cardiac-ischemia/infarction (Cardiac disorders) | 0 | 1 — Grade 4
Bradycardia and dyspnea (Cardiac disorders) | 0 | 1 — Grade 2
Septic shock (Infections and infestations) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 — Grade 2
SGOT (AST) and SGPT (ALT) (Hepatobiliary disorders) | 0 | 1 — Grade 4
Leukocytes (Blood and lymphatic system disorders) | 1 | 0 — Grade 4 and Fever grade 1
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1 — Grade 3
Fatigue (General disorders) | 0 | 2 — Grade 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: FAC (N=974) | Arm B: FAC-wP (N=951)
Neutrophils/Granulocytes (Blood and lymphatic system disorders) | 250 | 203 — Grade 3-4
Febrile neutropenia (General disorders) | 36 | 25 — Grade 3-4
Infection without neutropenia (Infections and infestations) | 3 | 13 — Grade 3-4
Infection with unknown ANC (Infections and infestations) | 3 | 11 — Grade 3-4
Lymphopenia (Blood and lymphatic system disorders) | 10 | 8 — Grade 3-4
Leukocytes (Blood and lymphatic system disorders) | 93 | 78 — Grade 3-4
SGPT (ALT) (Investigations) | 10 | 22 — Grade 3-4
Irregular Menses (Reproductive system and breast disorders) | 105 | 148 — Grade 3-4
Fatigue (General disorders) | 34 | 74 — Grade 3-4
Neurophaty-sensory (Nervous system disorders) | 0 | 51 — Grade 3-4
Vomiting (Gastrointestinal disorders) | 40 | 40 — Grade 3-4
Nausea (Gastrointestinal disorders) | 25 | 25 — Grade 3-4
STOMATITIS/PHARYNGITIS (ORAL/PHARYNGEAL MUCOSITIS) (Gastrointestinal disorders) | 17 | 16 — Grade 3-4
Myalgia (Nervous system disorders) | 2 | 14 — Grade 3-4
CNS cerebrovascular ischemia (Nervous system disorders) | 1 | 0 — Grade 3-4
Thrombosis/embolism (Cardiac disorders) | 1 | 10 — Grade 3-4
Cardiac Function (Cardiac disorders) | 0 | 1 — Grade 3-4
Cardiac Left Ventricular (Cardiac disorders) | 0 | 1 — Grade 3-4
Cardiac-ischemia/infarction (Cardiac disorders) | 1 | 1 — Grade 3-4
DIARRHEA (Gastrointestinal disorders) | 3 | 9 — Grade 3-4
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 2 | 9 — Grade 3-4
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 7 — Grade 3-4
CONJUNCTIVITIS (Eye disorders) | 5 | 4 — Grade 3-4
CONSTIPATION (Gastrointestinal disorders) | 5 | 6 — Grade 3-4
GGT (Hepatobiliary disorders) | 3 | 5 — Grade 3-4
INFECTION WITH NEUTROPENIA (Infections and infestations) | 9 | 6 — Grade 3-4
PLATELETS (Blood and lymphatic system disorders) | 5 | 3 — Grade 3-4
SGOT (AST) (Hepatobiliary disorders) | 4 | 7 — Grade 3-4
ALLERGIC REACTION/HYPERSENSITIVITY (Immune system disorders) | 0 | 3 — Grade 3-4
BONE PAIN (Investigations) | 2 | 3 — Grade 3-4
HEMOGLOBIN (Blood and lymphatic system disorders) | 4 | 6 — Grade 3-4
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 0 | 5 — Grade 3-4
MUCOSITIS (Gastrointestinal disorders) | 4 | 2 — Grade 3-4
MOOD ALTERATION-ANXIETY, AGITATION (Nervous system disorders) | 1 | 4 — Grade 3-4
HAND FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 0 | 5 — Grade 3-4
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 4 | 2 — Grade 3-4
DYSPEPSIA/HEARTBURN (Gastrointestinal disorders) | 3 | 1 — Grade 3-4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 9 — Grade 3-4
ANOREXIA (Gastrointestinal disorders) | 0 | 2 — Grade 3-4
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 2 — Grade 3-4
PNEUMONITIS/PULMONARY INFILTRATES (Infections and infestations) | 0 | 2 — Grade 3-4
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 2 — Grade 3-4
PULMONARY (Respiratory, thoracic and mediastinal disorders) | 0 | 2 — Grade 3-4
SYNCOPE (FAINTING) (Cardiac disorders) | 2 | 1 — Grade 3-4
VASOVAGAL EPISODE (Cardiac disorders) | 1 | 3 — Grade 3-4
WEIGHT GAIN (General disorders) | 1 | 6 — Grade 3-4
WEIGHT LOSS (General disorders) | 2 | 1 — Grade 3-4
BILIRUBIN (Blood and lymphatic system disorders) | 1 | 1 — Grade 3-4
HOT FLASHES/FLUSHES (Reproductive system and breast disorders) | 1 | 1 — Grade 3-4
INFECTION (Infections and infestations) | 1 | 1 — Grade 3-4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less